CLINICAL TRIAL: NCT01853761
Title: Microcurrent and Aerobic Exercise Effects on Abdominal Fat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Escola Superior de Tecnologia da Saúde do Porto (Other)
Responsible Party: Principal Investigator, Andreia Noites, Professor, Escola Superior de Tecnologia da Saúde do Porto
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: AN-001
Record Dates: First submitted 2013-04-18; First posted 2013-05-15 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2013-05

CONDITIONS: Obesity, Abdominal
Keywords: abdominal fat; metabolic syndrome; microcurrent; aerobic exercise
MeSH Terms: conditions — Obesity, Abdominal; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Exercise after, Transcutaneos, 25-10Hz (Experimental): Experimental group 1 performed aerobic exercise just after microcurrent in the abdominal region with four transcutaneous electrodes in a parallel position, intensity below the sensivity threshold and a maximum of 1 mA. Every 15 minutes changed from 25Hz to 10 Hz.
  Interventions: Device: Exercise after; Device: Transcutaneos; Device: 25-10Hz
- 25-50Hz microcurrent (Experimental): Experimental group 2 performed aerobic exercise just after microcurrent in the abdominal region with four transcutaneous electrodes in a parallel position, intensity below the sensivity threshold and a maximum of 1 mA. Every 15 minutes changed from 25Hz to 50Hz.
  Interventions: Device: Exercise after; Device: Transcutaneos; Device: 25-50Hz microcurrent
- percutaneous microcurrent (Experimental): Experimental group 3 performed aerobic exercise just after microcurrent in the abdominal region with four percutaneous electrodes in a parallel position, intensity below the sensivity threshold and a maximum of 1 mA. Every 15 minutes changed from 25Hz to 10 Hz.
  Interventions: Device: Exercise after; Device: percutaneous microcurrent; Device: 25-10Hz
- Exercise at same time (Experimental): Experimental group 4 performed aerobic exercise at the same time microcurrent in the abdominal region with four transcutaneous electrodes in a parallel position, intensity below the sensivity threshold and a maximum of 1 mA. Every 15 minutes changed from 25Hz to 10 Hz.
  Interventions: Device: Exercise at same time; Device: Transcutaneos; Device: 25-10Hz
- Control Group (Placebo Comparator): Control group performed aerobic exercise just after microcurrent in the abdominal region with four transcutaneous electrodes in a parallel position, but microcurrent device was switched off.
  Interventions: Device: Exercise after; Device: Transcutaneos

INTERVENTIONS:
Device: Exercise after — Aerobic exercise just after microcurrent in the abdominal region, intensity below the sensivity threshold and a maximum of 1 mA.
  30 minutes of aerobic moderate-intensity exercise (50%VO2 max) using Karvonen´s formula, performed on a cycloergometer. Were used Borg scale (12-13) and Polar® heart monitors to control heart rate.
  Other Names: Aerobic exercise after microcurrent
  Arms: 25-50Hz microcurrent; Control Group; Exercise after, Transcutaneos, 25-10Hz; percutaneous microcurrent
Device: Exercise at same time — Aerobic exercise at the same time microcurrent in the abdominal region, intensity below the sensivity threshold and a maximum of 1 mA.
  30 minutes of aerobic moderate-intensity exercise (50%VO2 max) using Karvonen´s formula, performed on a cycloergometer. Were used Borg scale (12-13) and Polar® heart monitors to control heart rate.
  Other Names: Aerobic exercise at same time microcurrent
  Arms: Exercise at same time
Device: Transcutaneos — Microcurrent device in the abdominal region with four transcutaneous electrodes in a parallel position, intensity below the sensivity threshold and a maximum of 1 mA.
  Other Names: transcutaneos microcurrent
  Arms: 25-50Hz microcurrent; Control Group; Exercise after, Transcutaneos, 25-10Hz; Exercise at same time
Device: percutaneous microcurrent — Microcurrent device in the abdominal region with four percutaneous electrodes in a parallel position, intensity below the sensivity threshold and a maximum of 1 mA.
  Arms: percutaneous microcurrent
Device: 25-10Hz — microcurrent device in the abdominal whith intensity below the sensivity threshold and a maximum of 1 mA. Every 15 minutes changed from 25Hz to 10 Hz.
  Other Names: 25-10Hz microcurrent
  Arms: Exercise after, Transcutaneos, 25-10Hz; Exercise at same time; percutaneous microcurrent
Device: 25-50Hz microcurrent — microcurrent device in the abdominal whith intensity below the sensivity threshold and a maximum of 1 mA. Every 15 minutes changed from 25Hz to 50 Hz.
  Arms: 25-50Hz microcurrent

SUMMARY:
The purpose of this study was to analyze microcurrent short and long term effects used with aerobic exercise on abdominal fat.

DETAILED DESCRIPTION:
Nutritional patterns have been changed during XXI century with sugar and fat's high proportions that allied to sedentarism increased body fat. There is already a well establish relationship between total body fat excess, cardiometabolic diseases and increased mortality, knowing that abdominal fat (android pattern), different from body index, presents an additional influence to health risks. Women with their abdominal adipocytes (visceral fat) show an increased lipolitic activity that releases free fat acids to the systemic and portal circulation leading to a metabolic syndrome, increasing the risk of cardiovascular diseases Aerobic exercise is a way to decrease fat as it stimulates lipolysis through an increase in catecholamine's level resulting from a sympathetic system nervous activity raise. The most used exercise for lipid elimination is the prolonged aerobic moderate exercise with a minimum of 30 mn.

Nevertheless aerobic exercise practice reduce globally lipidic sources and not locally . Electrolipolysis using microcurrent has been used in clinical practice as a technique to reduce abdominal fat. This technique can be applied transcutaneously or percutaneously seeming that the former is not so effective as skin can be an obstacle to the current effect on visceral and subcutaneous fat .

Abdominal fat excess is associated with cardiometabolic diseases and can be prevented using microcurrent and aerobic exercise to stimulate lipolysis.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 30 years
* presenting a normal to pre-obese body mass index (18.5 - 29.9 Kg/m2)
* moderate physical activity level (between 600 and 3000 metabolic-minute/week (MET-min/week)) scored by International Physical Activity Questionnaire (IPAQ)

Exclusion Criteria:

* submitted to other fat reduce procedure
* to show cardiovascular risk factors or diseases and/or any physical condition limiting aerobic exercise
* to present any contra indications to microcurrent and/or aerobic exercise
* to take medication that influence lipid metabolism, and to be pregnant

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2011-07; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
subcutaneous abdominal fat and viceral abdominal fat | five weeks after the intervencion
  Ultrasound was performed at the end of expiration to measure subcutaneous abdominal fat between xiphoid apophysis and navel, below navel, and above left and right anterior superior iliac spine. Between xiphoid apophysis and navel was also measured visceral abdominal fat

SECONDARY OUTCOMES:
bioimpedance values | five weeks after the intervencion
  The height was measured with the volunteers on respiratory apnea. To minimize the influence of electrolyte balance changes in bioimpedance assessment, was given some rules to volunteers. It was calculated BMI using the body weight divided by height squared.
cholesterol, triglycerides and glucose levels | five weeks after intervention
  The volunteers were on fasting (12 hours) and was collected a blood sample on finger to measure cholesterol, triglycerides and glucose levels. The results were recorded through the classes
perimeters measurements | five weeks after intervencion
  The perimeters measurements were done, at the end of expiration, at waist level (below last rib), at navel level, at the point immediately above the iliac crests and at trochanters level. The waist-hip ratio was calculated using the waist level perimeter divided by trochanters level perimeter
Suprailiac, vertical and horizontal abdominal skinfolds | five weeks after intervencion
  Suprailiac, vertical and horizontal abdominal skinfolds were performed three times in right hemi body, by caliper

OTHER OUTCOMES:
International Physical Activity Questionnaire | five weeks after the intervencion
  moderate physical activity level were used to monitor lifestyle during sessions
Food Frequency Questionnaire | five weeks after intervencion
  Food Frequency Questionnaire were used to monitor lifestyle during sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Andreia Noites, MSc, Principal Investigator — Escola Superior de Tecnologia da Saúde do Porto
Locations (1):
- Andreia Noites, Vila Nova de Gaia, Porto District, Portugal

REFERENCES:
- [Background] Despres JP, Lemieux I. Abdominal obesity and metabolic syndrome. Nature. 2006 Dec 14;444(7121):881-7. doi: 10.1038/nature05488. PMID 17167477
- [Background] Donnelly JE, Blair SN, Jakicic JM, Manore MM, Rankin JW, Smith BK; American College of Sports Medicine. American College of Sports Medicine Position Stand. Appropriate physical activity intervention strategies for weight loss and prevention of weight regain for adults. Med Sci Sports Exerc. 2009 Feb;41(2):459-71. doi: 10.1249/MSS.0b013e3181949333. PMID 19127177
- [Background] Ribeiro-Filho FF, Faria AN, Azjen S, Zanella MT, Ferreira SR. Methods of estimation of visceral fat: advantages of ultrasonography. Obes Res. 2003 Dec;11(12):1488-94. doi: 10.1038/oby.2003.199. PMID 14694213
- [Background] Hamida ZH, Comtois AS, Portmann M, Boucher JP, Savard R. Effect of electrical stimulation on lipolysis of human white adipocytes. Appl Physiol Nutr Metab. 2011 Apr;36(2):271-5. doi: 10.1139/h11-011. PMID 21609289